CLINICAL TRIAL: NCT04986540
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Dose Escalation Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of Single IV Infusion of SHR-1906 in Healthy Subjects
Brief Title: A Trial of SHR - 1906 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guangdong Hengrui Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1906-101
Record Dates: First submitted 2021-07-27; First posted 2021-08-03 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Idiopathic Pulmonary Fibrosis
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Intervention Model Description: SHR-1906 compared with placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1 (Experimental): A single subcutaneous injection of SHR-1906/placebo dose 1 in healthy subjects
  Interventions: Drug: SHR-1906；Placebo
- Cohort 2 (Experimental): A single subcutaneous injection of SHR-1906/placebo dose 2 in healthy subjects
  Interventions: Drug: SHR-1906；Placebo
- Cohort 3 (Experimental): A single subcutaneous injection of SHR-1906/placebo dose 3 in healthy subjects
  Interventions: Drug: SHR-1906；Placebo
- Cohort 4 (Experimental): A single subcutaneous injection of SHR-1906/placebo dose 4 in healthy subjects
  Interventions: Drug: SHR-1906；Placebo
- Cohort 5 (Experimental): A single subcutaneous injection of SHR-1906/placebo dose 5 in healthy subjects
  Interventions: Drug: SHR-1906；Placebo
- Cohort 6 (Experimental): A single subcutaneous injection of SHR-1906/placebo dose 6 in healthy subjects
  Interventions: Drug: SHR-1906；Placebo

INTERVENTIONS:
Drug: SHR-1906；Placebo — Drug: SHR-1906 IV, single dose
  Drug: Placebo IV, single dose

SUMMARY:
This study is a phase 1 single dose escalation study of SHR-1906 in healthy subjects. The purpose of the study is to evaluate the safety, tolerability and pharmacokinetics of SHR-1906 in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand the trial procedures and possible adverse events, volunteers to participate in the trial, and provides written informed consent, be able to comply with all the requirements and able to complete the study.
2. Male or female aged between 18 years and 55 years (inclusive) at the date of signed consent form.
3. Total body weight ≥ 45 kg.
4. No clinically significant abnormalities in medical history, general physical examination, vital signs, laboratory tests (hematology, urinalysis, blood chemistry, coagulation function and thyroid function) and ECG at the investigator's discretion during screening and baseline
5. Men and women of childbearing potential (WOCBP) must agree to take effective contraceptive methods

Exclusion Criteria:

1. History of serious cardiovascular, liver, kidney, digestive tract, psychiatric, hematology, metabolic disorders, primary immunodeficiency disease or acquired immune deficiency syndrome, or organ transplantation.
2. Severe infections, injuries or major surgeries (as determined by the investigator) within 6 months prior to screening, or plan to do any surgery during the trial.
3. Positive testing for human immunodeficiency virus (HIV-Ab), or hepatitis B surface antigen (HBsAg), or TP-Ab , or hepatitis C antibodies (HCV-Ab).
4. Screening/baseline systolic blood pressure (BP) ≥140 mmHg or ≤90 mmHg; diastolic BP ≥90 mmHg or <60 mmHg on a single measurement
5. Positive urine drug screening at baseline;
6. Use of any medicine within 1 monthes (including any prescription, or over-the-counter medicine, herbal remedy or nutritional supplement, except for vitamins and occasional use of acetaminophen with recommended dose), or within 5 half-lives of any drugs whichever is longer prior to dosing, or plan to use any medicine during the trial.
7. Participation in clinical trials of other investigational drugs or medical devices within 3 months prior to screening or within 5 half-lives of any drugs during screening visit, or in the follow-up period of a clinical study whichever is longer (according to the date of signed consent form) which is defined as having consented and used other investigational drugs (including placebo) or trial medical devices.
8. Blood donation or loss of ≥ 400 mL of blood within 1 months; or received blood or blood products within 2 months prior to screening.
9. Any other circumstances that, in the investigator's judgment, may increase the risk associated with the subject's participation in and completion of the study or could preclude the evaluation of the subject's response.
10. Researchers and relevant staff of the research center or other persons directly involved in the implementation of the program.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2021-08-10 (Actual); Primary Completion 2022-09-07 (Actual); Study Completion 2022-09-07 (Actual)

PRIMARY OUTCOMES:
Adverse events | Start of Treatment to end of study (approximately 10 weeks)
  Incidence and severity of adverse events

SECONDARY OUTCOMES:
Pharmacokinetics-AUC0-last | Start of Treatment to end of study (approximately 10 weeks)
  Area under the concentration-time curve from time 0 to last time point after SHR-1906 administration
Pharmacokinetics-AUC0-inf | Start of Treatment to end of study (approximately 10 weeks)
  Area under the concentration-time curve from time 0 to infinity after SHR-1906 administration
Pharmacokinetics-Tmax | Start of Treatment to end of study (approximately 10 weeks)
  Time to Cmax of SHR-1906
Pharmacokinetics-Cmax | Start of Treatment to end of study (approximately 10 weeks)
  Maximum observed concentration of SHR-1906
Pharmacokinetics-CL | Start of Treatment to end of study (approximately 10 weeks)
  Clearance of SHR-1906
Pharmacokinetics-V | Start of Treatment to end of study (approximately 10 weeks)
  Volume of distribution during terminal phase of SHR-1906
Pharmacokinetics-t1/2 | Start of Treatment to end of study (approximately 10 weeks)
  Terminal elimination half-life of SHR-1906
Anti-Drug antibody | Start of Treatment to end of study (approximately 10 weeks)
  The percentage of subjects with positive ADA titers over time for SHR-1906

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Clinical Research Unit, Qianfoshan Hospital of Shandong Province, Jinan, Shandong, China